CLINICAL TRIAL: NCT01595009
Title: An Open-label, Multi-center, Expanded Access Study of Everolimus in Participants With Advanced Neuroendocrine Tumors (NETs) (Core Study) and an Extension Study to the Open-label, Multi-center, Expanded Access Study of Everolimus in Patients With Advanced NETs (E1)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001K24133
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (RAD001) (Experimental): Participants received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001) — Everolimus was supplied as tablets of 5mg strength.
  Other Names: Afinitor

SUMMARY:
This record combines the results of CRAD001K24133 and CRAD001K24133E1. The purpose of the CRAD001K24133 study was to evaluate the safety profile of everolimus in patients with advanced neuroendocrine tumors of pancreatic origin (pNETs) and to provide access of everolimus to this patient population. Everolimus was taken by participants until disease progression, unacceptable toxicity, death, discontinuation from the trial for any other reason, or when it became commercially available for this indication, or until May 30, 2012, whichever came first. Prior to amendment 1, the study enrolled participants with NET of the lung (L-NETs) and gastrointestinal (GI) (GI-NETs) origin. The core study was stopped (per protocol) because everolimus was approved for pNETs. All ongoing patients with pNETs were switched to commercially available everolimus. For GI and lung NETs, everolimus was not approved at the time the core study was stopped. Therefore, patients with GI or lung NETs were not able to switch to commercial drug. To provide study medication access to these patients beyond 30 May 2012, the open label extension study, CRAD001K24133E1, was conducted. In the extension study, RAD001K24133E1, participants with GI or lung NETs who had not progressed during therapy with everolimus in the core study and who had not suffered from intolerable toxicity, were enrolled and treated with everolimus in order to provide data on long-term safety and efficacy. Patients were treated until it became commercially available in the respective indication or until documented tumor progression, unacceptable toxicity, any other reason or until study end on 31 May 2017, whichever came first.

ELIGIBILITY:
Core Inclusion:

* Age ≥ 18 years old
* Advanced (unresectable or metastatic) biopsy-proven NETs of pancreatic origin
* World health organization (WHO) Performance status of 0-2
* Adequate bone marrow function as shown by:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin >9 g/dL
* Adequate liver function as shown by:
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN. Patients with known liver metastases with an AST and ALT ≤ 5 x ULN
* International normalized ratio (INR) <1.3 (INR <3 in patients treated with anticoagulants)
* Adequate renal function as shown by: Serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤ 300 mg/dL or ≤ 7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN
* Written informed consent obtained before any trial related activity and according to local guidelines.

Core Exclusion:

* Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid and small cell carcinoma were not eligible.
* Following Amendment 1, patients with neuroendocrine tumors of GI or lung origin
* Cytotoxic chemotherapy, immunotherapy or radiotherapy within 4 weeks prior to enrollment
* Hepatic artery embolization within the last two months or cryoablation or radiofrequency ablation of hepatic metastasis within two months of enrollment
* Prior therapy with mTOR inhibitors (for example sirolimus, temsirolimus, everolimus)
* Patients with a known hypersensitivity to everolimus or other rapamycin analogs (sirolimus, temsirolimus) or to its excipients
* Patients receiving chronic treatment with immunosuppressives
* Uncontrolled diabetes mellitus as defined by fasting serum glucose >1.5 x ULN
* Patients who had any severe and/or uncontrolled medical conditions such as:

Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction

≤ 6 months prior to enrollment, serious uncontrolled cardiac arrhythmia

* Active or uncontrolled severe infection
* A history of invasive fungal infections
* Severe hepatic impairment (Child Pugh class C)
* Severely impaired lung function
* Active bleeding diathesis
* Patients with a known history of Human immunodeficiency virus (HIV) seropositivity
* No other prior or concurrent malignancy was allowed except for, adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient had been disease free for ≥ 3 years
* Patients within four weeks post-major surgery, open-biopsy, or significant traumatic injury to avoid wound healing complications. Minor procedures and percutaneous biopsies or placement of vascular access device required seven days prior to study entry
* Female patients who were pregnant or nursing
* Adults who were of reproductive potential who were not using effective birth control methods. Adequate contraceptives were to be used throughout the trial and for eight weeks after last study drug administration in female patients. Women of child bearing potential must have had a negative serum pregnancy test within seven days prior to first administration of study drug
* Patients who were unwilling to or unable to comply with the protocol

Extension Inclusion and Exclusion Criteria:

* The patient must provide a signed Informed Consent Form (ICF) for the extension study prior to any study related procedures
* Age ≥18 years old
* Completion of the whole treatment period in the CRAD001K24133 study
* Neuroendocrine tumor of gastrointestinal or pulmonary origin (pancreatic neuroendocrine tumors are excluded)
* No tumor progression during therapy with everolimus during CRAD001K24133 study (checked via radiologically assessment)
* No intolerable toxicity during therapy everolimus, or during combination therapy of everolimus and somatostatin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2011-04-27; Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Weiden

RESULTS

PARTICIPANT FLOW:
Groups:
- pNET (Core): Participants with NETs of a pancreatic origin received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
- Non-pNET (Core): Participants with NETs of a GI or lung origin received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
- Lung NET (E1): Participants with NETs of a lung origin received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
- GI NET (E1): Participants with NETs of a GI origin received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
Period: Core
Arm/Group | pNET (Core) | Non-pNET (Core) | Lung NET (E1) | GI NET (E1)
Started | 126 | 120 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 126 | 120 | 0 | 0
Not completed — Patients completed per protocol | 85 | 44 | 0 | 0
Not completed — Adverse Event | 19 | 23 | 0 | 0
Not completed — Disease progression | 14 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 17 | 0 | 0
Not completed — Death | 3 | 6 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0
Not completed — Administrative problems | 0 | 1 | 0 | 0
Period: Extension
Arm/Group | pNET (Core) | Non-pNET (Core) | Lung NET (E1) | GI NET (E1)
Started | 0 | 0 | 4 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 4 | 11
Not completed — Administrative problems | 0 | 0 | 0 | 1
Not completed — Patients completed per protocol | 0 | 0 | 0 | 2
Not completed — Disease progression | 0 | 0 | 4 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | pNET (Core) | Non-pNET (Core) | Total
Number analyzed (Participants) | 126 | 120 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.04) | 64.4 (9.28) | 61.8 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 119
  Male | 68 | 59 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths (Core)
Description: The number of participants with AEs, SAEs and deaths were assessed.
Time Frame: from the day of first treatment up to 19 months
Population: The safety population, which consisted of all patients who received at least one dose of everolimus and had at least one post-baseline safety assessment, was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 123 | 117
Participants
  Adverse events | 90 | 109
  Serious adverse events | 25 | 59
  Deaths | 5 | 10

2. Primary Outcome: Number and Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths During the Extension Phase (E1)
Description: The number of participants with AEs, SAEs and deaths were assessed.
Time Frame: from the first day of treatment in the extension up to 4 years
Population: The safety set, which consisted of all participants who received at least one dose of everolimus during the extension and had at least one post-baseline safety assessment during the extension, was analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- GI NET: Participants with NETs of a GI origin received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
Arm/Group | Lung NET (E1) | GI NET
Number analyzed (Participants) | 4 | 11
Participants
  AEs | 4 | 11
  SAEs | 1 | 4
  Deaths | 0 | 1

3. Secondary Outcome: Investigator-assessed Progression Free Survival (PFS) (Core)
Description: PFS was defined as the time from the date of the first dose to the date of the first radiologically documented disease progression or death due to any cause. If a participant had not progressed or died at the study end date or when he/she received any further anti-neoplastic therapy, PFS was censored at the time of the last tumor assessment before the end of study date. Progression was defined,using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from the day of first treatment up to 19 months
Population: The full analysis set, which consisted of all participants who received at least one dose, was analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 126 | 120
Months | 7.62 [5.52 to 7.62] | 10.78 [8.77 to NA] — Upper limit of the 95% confidence interval was not estimable because there were too few participants at this time point.

4. Secondary Outcome: Mean European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) Score (Core)
Description: The EORTC QLQ-C30 contains 30 questions assessed by the participant. There are 9 multiple-item scales: 5 scales that assess aspects of functioning (physical, role functioning, cognitive, emotional, and social); 3 symptom scales (Fatigue, Pain, and Nausea and Vomiting); and a global health status/Quality of Life (QOL) scale. There are 5 single-item measures assessing additional symptoms (i.e., dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and a single item concerning perceived financial impact of the disease. All but two questions have 4-point scales ranging from "Not at all" to "Very much." The two questions concerning global health status/ QOL have 7 point scales with ratings ranging from "Very poor" to "Excellent." For each of the 14 domains, final scores are transformed such that they range from 0-100, where higher scores indicate improvement.
Time Frame: Baseline, weeks 4, 8, 20, 32, 44, and end of treatment (EOT) up to week 82
Population: The full analysis set, which consisted of all participants who received at least one dose of everolimus, was considered for the analysis. Only participants with measurement at each given time point were analyzed for that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 126 | 120
units on a scale
  Global health status/QOL, Baseline: number analyzed (Participants) | 120 | 110
  Global health status/QOL, Baseline | 64.93 (20.946) | 60.53 (21.497)
  Global health status/QOL, Week 4: number analyzed (Participants) | 102 | 102
  Global health status/QOL, Week 4 | 63.15 (19.673) | 58.91 (20.622)
  Global health status/QOL, Week 8: number analyzed (Participants) | 72 | 86
  Global health status/QOL, Week 8 | 59.72 (21.303) | 56.59 (20.417)
  Global health status/QOL,Week 20: number analyzed (Participants) | 28 | 57
  Global health status/QOL,Week 20 | 63.10 (22.387) | 59.65 (17.663)
  Global health status/QOL, Week 32: number analyzed (Participants) | 5 | 39
  Global health status/QOL, Week 32 | 50.0 (26.352) | 56.20 (20.297)
  Global health status/QOL, Week 44: number analyzed (Participants) | 3 | 14
  Global health status/QOL, Week 44 | 61.11 (9.623) | 57.74 (25.205)
  Global health status/QOL, EOT up to Week 82: number analyzed (Participants) | 87 | 73
  Global health status/QOL, EOT up to Week 82 | 61.40 (20.847) | 48.86 (27.823)
  Physical functioning, Baseline: number analyzed (Participants) | 120 | 111
  Physical functioning, Baseline | 79.89 (20.850) | 72.97 (22.938)
  Physical functioning, week 4: number analyzed (Participants) | 103 | 103
  Physical functioning, week 4 | 77.02 (22.380) | 68.62 (23.648)
  Physical functioning, week 8: number analyzed (Participants) | 74 | 88
  Physical functioning, week 8 | 76.22 (25.810) | 67.48 (24.973)
  Physical functioning, week 20: number analyzed (Participants) | 29 | 57
  Physical functioning, week 20 | 79.77 (18.212) | 73.71 (21.351)
  Physical functioning, week 32: number analyzed (Participants) | 5 | 39
  Physical functioning, week 32 | 68.00 (26.415) | 71.62 (23.729)
  Physical functioning, week 44: number analyzed (Participants) | 3 | 14
  Physical functioning, week 44 | 68.89 (13.878) | 76.19 (22.602)
  Physical functioning, EOT up to week 82: number analyzed (Participants) | 86 | 76
  Physical functioning, EOT up to week 82 | 75.70 (24.509) | 60.94 (28.037)
  Role functioning, Baseline: number analyzed (Participants) | 120 | 110
  Role functioning, Baseline | 75.28 (28.663) | 67.27 (32.397)
  Role functioning, week 4: number analyzed (Participants) | 103 | 102
  Role functioning, week 4 | 72.49 (28.364) | 62.25 (30.483)
  Role functioning, week 8: number analyzed (Participants) | 71 | 88
  Role functioning, week 8 | 71.83 (30.025) | 58.14 (31.460)
  Role functioning, week 20: number analyzed (Participants) | 28 | 56
  Role functioning, week 20 | 79.76 (25.803) | 58.33 (29.129)
  Role functioning, week 32: number analyzed (Participants) | 5 | 38
  Role functioning, week 32 | 66.67 (26.352) | 55.26 (35.325)
  Role functioning, week 44: number analyzed (Participants) | 3 | 14
  Role functioning, week 44 | 61.11 (9.623) | 66.67 (26.954)
  Role functioning, EOT up to week 82: number analyzed (Participants) | 85 | 77
  Role functioning, EOT up to week 82 | 67.84 (31.788) | 49.13 (33.212)
  Emotional functioning, Baseline: number analyzed (Participants) | 120 | 110
  Emotional functioning, Baseline | 74.79 (22.650) | 67.20 (22.988)
  Emotional functioning, week 4: number analyzed (Participants) | 102 | 103
  Emotional functioning, week 4 | 76.31 (20.991) | 66.69 (25.380)
  Emotional functioning, week 8: number analyzed (Participants) | 72 | 88
  Emotional functioning, week 8 | 73.38 (24.730) | 64.02 (26.640)
  Emotional functioning, week 20: number analyzed (Participants) | 28 | 57
  Emotional functioning, week 20 | 76.19 (19.072) | 63.16 (27.456)
  Emotional functioning, week 32: number analyzed (Participants) | 5 | 39
  Emotional functioning, week 32 | 81.67 (14.907) | 61.11 (28.184)
  Emotional functioning, week 44: number analyzed (Participants) | 3 | 14
  Emotional functioning, week 44 | 75.00 (8.333) | 65.67 (31.059)
  Emotional functioning, EOT up to week 82: number analyzed (Participants) | 86 | 75
  Emotional functioning, EOT up to week 82 | 74.61 (23.602) | 57.63 (25.841)
  Cognitive functioning, Baseline: number analyzed (Participants) | 119 | 110
  Cognitive functioning, Baseline | 84.17 (19.630) | 80.61 (23.842)
  Cognitive functioning, week 4: number analyzed (Participants) | 102 | 103
  Cognitive functioning, week 4 | 86.11 (20.050) | 78.80 (23.708)
  Cognitive functioning, week 8: number analyzed (Participants) | 72 | 88
  Cognitive functioning, week 8 | 81.94 (21.803) | 76.33 (27.418)
  Cognitive functioning, week 20: number analyzed (Participants) | 28 | 57
  Cognitive functioning, week 20 | 83.93 (19.501) | 78.65 (23.307)
  Cognitive functioning, week 32: number analyzed (Participants) | 5 | 39
  Cognitive functioning, week 32 | 86.67 (18.257) | 75.21 (24.445)
  Cognitive functioning, week 44: number analyzed (Participants) | 3 | 14
  Cognitive functioning, week 44 | 94.44 (9.623) | 84.52 (20.111)
  Cognitive functioning, EOT up to week 82: number analyzed (Participants) | 84 | 76
  Cognitive functioning, EOT up to week 82 | 81.35 (21.241) | 73.46 (24.522)
  Social functioning, Baseline: number analyzed (Participants) | 120 | 111
  Social functioning, Baseline | 75.56 (28.249) | 67.42 (28.989)
  Social functioning, week 4: number analyzed (Participants) | 101 | 103
  Social functioning, week 4 | 78.71 (23.347) | 67.80 (30.093)
  Social functioning, week 8: number analyzed (Participants) | 72 | 86
  Social functioning, week 8 | 75.69 (24.695) | 65.31 (29.396)
  Social functioning, week 20: number analyzed (Participants) | 28 | 56
  Social functioning, week 20 | 73.21 (24.148) | 66.07 (29.977)
  Social functioning, week 32: number analyzed (Participants) | 5 | 39
  Social functioning, week 32 | 60.00 (27.889) | 66.24 (32.329)
  Social functioning, week 44: number analyzed (Participants) | 3 | 14
  Social functioning, week 44 | 66.67 (0.000) | 72.62 (31.082)
  Social functioning, EOT up to week 82: number analyzed (Participants) | 85 | 75
  Social functioning, EOT up to week 82 | 75.10 (27.533) | 52.89 (33.933)
  Fatigue, baseline: number analyzed (Participants) | 120 | 111
  Fatigue, baseline | 31.30 (22.361) | 42.39 (28.534)
  Fatigue, week 4: number analyzed (Participants) | 103 | 103
  Fatigue, week 4 | 35.22 (22.887) | 43.58 (28.035)
  Fatigue, week 8: number analyzed (Participants) | 73 | 88
  Fatigue, week 8 | 36.91 (25.515) | 48.86 (29.878)
  Fatigue, week 20: number analyzed (Participants) | 29 | 57
  Fatigue, week 20 | 34.29 (18.430) | 44.44 (27.698)
  Fatigue, week 32: number analyzed (Participants) | 5 | 39
  Fatigue, week 32 | 42.22 (18.257) | 48.72 (29.575)
  Fatigue, week 44: number analyzed (Participants) | 3 | 14
  Fatigue, week 44 | 37.04 (6.415) | 38.89 (26.777)
  Fatigue, EOT up to week 82: number analyzed (Participants) | 87 | 77
  Fatigue, EOT up to week 82 | 38.83 (24.896) | 56.49 (30.474)
  Nausea and vomiting, Baseline: number analyzed (Participants) | 120 | 111
  Nausea and vomiting, Baseline | 11.25 (17.442) | 9.46 (17.353)
  Nausea and vomiting, week 4: number analyzed (Participants) | 103 | 101
  Nausea and vomiting, week 4 | 10.52 (15.998) | 7.43 (14.995)
  Nausea and vomiting, week 8: number analyzed (Participants) | 73 | 87
  Nausea and vomiting, week 8 | 9.59 (17.984) | 10.34 (18.015)
  Nausea and vomiting, week 20: number analyzed (Participants) | 29 | 57
  Nausea and vomiting, week 20 | 8.05 (15.185) | 6.14 (12.048)
  Nausea and vomiting, week 32: number analyzed (Participants) | 5 | 39
  Nausea and vomiting, week 32 | 6.67 (9.129) | 5.98 (11.139)
  Nausea and vomiting, week 44: number analyzed (Participants) | 3 | 14
  Nausea and vomiting, week 44 | 11.11 (9.623) | 4.76 (10.187)
  Nausea and vomiting, EOT up to week 82: number analyzed (Participants) | 86 | 77
  Nausea and vomiting, EOT up to week 82 | 9.69 (17.048) | 15.80 (27.023)
  Pain, Baseline: number analyzed (Participants) | 119 | 110
  Pain, Baseline | 21.57 (24.582) | 31.21 (31.535)
  Pain, week 4: number analyzed (Participants) | 101 | 102
  Pain, week 4 | 25.91 (26.716) | 30.88 (29.796)
  Pain, week 8: number analyzed (Participants) | 72 | 87
  Pain, week 8 | 25.23 (27.972) | 37.55 (32.372)
  Pain, week 20: number analyzed (Participants) | 28 | 57
  Pain, week 20 | 27.98 (22.247) | 33.33 (32.581)
  Pain, week 32: number analyzed (Participants) | 5 | 39
  Pain, week 32 | 43.33 (27.889) | 34.62 (32.977)
  Pain, week 44: number analyzed (Participants) | 3 | 14
  Pain, week 44 | 38.89 (9.623) | 26.19 (30.462)
  Pain, EOT up to week 82: number analyzed (Participants) | 86 | 71
  Pain, EOT up to week 82 | 27.33 (28.343) | 43.90 (33.362)
  Dyspnea, Baseline: number analyzed (Participants) | 120 | 111
  Dyspnea, Baseline | 16.11 (22.448) | 24.32 (29.110)
  Dyspnea, week 4: number analyzed (Participants) | 103 | 102
  Dyspnea, week 4 | 17.80 (24.171) | 26.14 (28.388)
  Dyspnea, week 8: number analyzed (Participants) | 73 | 87
  Dyspnea, week 8 | 21.00 (27.502) | 29.12 (31.665)
  Dyspnea, week 20: number analyzed (Participants) | 29 | 57
  Dyspnea, week 20 | 11.49 (18.422) | 28.07 (30.072)
  Dyspnea, week 32: number analyzed (Participants) | 5 | 39
  Dyspnea, week 32 | 13.33 (18.257) | 35.90 (31.885)
  Dyspnea, week 44: number analyzed (Participants) | 3 | 14
  Dyspnea, week 44 | 22.22 (19.245) | 21.43 (28.063)
  Dyspnea, EOT up to week 82: number analyzed (Participants) | 86 | 77
  Dyspnea, EOT up to week 82 | 25.19 (30.222) | 33.77 (30.824)
  Insomnia, Baseline: number analyzed (Participants) | 120 | 110
  Insomnia, Baseline | 24.72 (30.093) | 28.18 (32.929)
  Insomnia, week 4: number analyzed (Participants) | 102 | 103
  Insomnia, week 4 | 27.78 (29.324) | 32.36 (30.769)
  Insomnia, week 8: number analyzed (Participants) | 73 | 85
  Insomnia, week 8 | 32.88 (30.171) | 29.02 (28.540)
  Insomnia, week 24: number analyzed (Participants) | 29 | 57
  Insomnia, week 24 | 24.14 (26.572) | 35.09 (32.380)
  Insomnia, week 32: number analyzed (Participants) | 5 | 38
  Insomnia, week 32 | 26.67 (27.889) | 33.33 (32.880)
  Insomnia, week 48: number analyzed (Participants) | 3 | 14
  Insomnia, week 48 | 22.22 (19.245) | 28.57 (36.648)
  Insomnia, EOT up o week 82: number analyzed (Participants) | 86 | 77
  Insomnia, EOT up o week 82 | 32.17 (31.289) | 34.63 (32.643)
  Appetite loss, Baseline: number analyzed (Participants) | 120 | 111
  Appetite loss, Baseline | 20.56 (30.613) | 18.62 (29.365)
  Appetitie loss, week 4: number analyzed (Participants) | 102 | 102
  Appetitie loss, week 4 | 25.16 (31.618) | 21.90 (29.849)
  Appetitie loss, week 8: number analyzed (Participants) | 73 | 87
  Appetitie loss, week 8 | 24.66 (30.946) | 25.67 (31.623)
  Appetitie loss, week 24: number analyzed (Participants) | 29 | 57
  Appetitie loss, week 24 | 18.39 (27.583) | 20.47 (27.998)
  Appetitie loss, week 36: number analyzed (Participants) | 5 | 39
  Appetitie loss, week 36 | 20.00 (18.257) | 23.93 (30.540)
  Appetitie loss, week 44: number analyzed (Participants) | 3 | 14
  Appetitie loss, week 44 | 11.11 (19.245) | 26.19 (29.753)
  Appetitie loss, EOT up to week 82: number analyzed (Participants) | 87 | 76
  Appetitie loss, EOT up to week 82 | 24.14 (29.505) | 33.77 (37.906)
  Constipation, Baseline: number analyzed (Participants) | 120 | 111
  Constipation, Baseline | 13.06 (24.175) | 13.21 (27.072)
  Constipation, week 4: number analyzed (Participants) | 103 | 103
  Constipation, week 4 | 11.00 (24.427) | 11.33 (24.501)
  Constipation, week 8: number analyzed (Participants) | 73 | 88
  Constipation, week 8 | 10.50 (24.137) | 7.58 (22.447)
  Constipation, week 20: number analyzed (Participants) | 29 | 57
  Constipation, week 20 | 6.90 (16.377) | 8.77 (21.387)
  Constipation, week 32: number analyzed (Participants) | 5 | 39
  Constipation, week 32 | 0.00 (0.000) | 4.27 (13.636)
  Constipation, week 44: number analyzed (Participants) | 3 | 14
  Constipation, week 44 | 0.00 (0.000) | 2.38 (8.909)
  Constipation, EOT up to week 82: number analyzed (Participants) | 86 | 77
  Constipation, EOT up to week 82 | 12.79 (24.611) | 10.39 (23.107)
  Diarrhea, Baseline: number analyzed (Participants) | 119 | 110
  Diarrhea, Baseline | 19.89 (29.535) | 36.67 (38.828)
  Diarrhea, week 4: number analyzed (Participants) | 102 | 103
  Diarrhea, week 4 | 20.92 (25.658) | 38.19 (36.577)
  Diarrhea, week 8: number analyzed (Participants) | 73 | 88
  Diarrhea, week 8 | 27.40 (29.576) | 42.42 (39.708)
  Diarrhea, week 20: number analyzed (Participants) | 28 | 57
  Diarrhea, week 20 | 16.67 (21.276) | 31.58 (29.828)
  Diarrhea, week 32: number analyzed (Participants) | 5 | 39
  Diarrhea, week 32 | 13.33 (18.257) | 40.17 (36.015)
  Diarrhea, week 44: number analyzed (Participants) | 3 | 14
  Diarrhea, week 44 | 22.22 (19.245) | 40.48 (37.390)
  Diarrhea, EOT up to week 82: number analyzed (Participants) | 86 | 76
  Diarrhea, EOT up to week 82 | 25.97 (32.095) | 39.04 (38.639)
  Financial difficulties, Baseline: number analyzed (Participants) | 119 | 111
  Financial difficulties, Baseline | 18.77 (26.975) | 16.52 (25.770)
  Financial difficulties, week 4: number analyzed (Participants) | 100 | 100
  Financial difficulties, week 4 | 16.67 (24.845) | 16.67 (27.010)
  Financial difficulties, week 8: number analyzed (Participants) | 72 | 87
  Financial difficulties, week 8 | 19.44 (26.091) | 16.86 (24.837)
  Financial difficulties, week 20: number analyzed (Participants) | 28 | 57
  Financial difficulties, week 20 | 21.43 (22.616) | 19.88 (27.357)
  Financial difficulties, week 32: number analyzed (Participants) | 5 | 39
  Financial difficulties, week 32 | 40.00 (27.889) | 21.37 (28.084)
  Financial difficulties, week 44: number analyzed (Participants) | 3 | 14
  Financial difficulties, week 44 | 22.22 (19.245) | 19.05 (25.198)
  Financial difficulties, EOT up to week 82: number analyzed (Participants) | 86 | 76
  Financial difficulties, EOT up to week 82 | 21.71 (27.897) | 27.63 (30.496)

5. Secondary Outcome: Mean EORTC QLQ-G.I. NET21 Score (Core)
Description: The EORTC QLQ-G.I. NET21 contains 21 questions and has three defined multi-item symptom scales (endocrine - 3 questions, gastrointestinal - 5 questions, and treatment related side effects - 3 questions), two single item symptoms (bone/muscle pain and concern about weight loss), two psychosocial scales (social function - 3 questions and disease-related worries - 3 questions) and two other single items (sexuality and communication). For each of the 9 domains, final scores are transformed such that they range from 0-100, where higher scores indicate worsening.
Time Frame: Baseline, weeks 4, 8, 20, 32, 44, and end of treatment (EOT) up to week 82
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 126 | 120
units on a scale
  Endocrine, Baseline: number analyzed (Participants) | 65 | 111
  Endocrine, Baseline | 12.99 (20.372) | 23.52 (23.771)
  Endocrine, week 4: number analyzed (Participants) | 53 | 99
  Endocrine, week 4 | 13.21 (17.440) | 17.85 (21.403)
  Endocrine, week 8: number analyzed (Participants) | 33 | 88
  Endocrine, week 8 | 13.47 (17.293) | 16.79 (20.216)
  Endocrine, week 20: number analyzed (Participants) | 8 | 56
  Endocrine, week 20 | 12.50 (12.511) | 15.87 (21.067)
  Endocrine, week 32: number analyzed (Participants) | 4 | 38
  Endocrine, week 32 | 16.67 (14.344) | 13.74 (17.978)
  Endocrine, week 44: number analyzed (Participants) | 1 | 14
  Endocrine, week 44 | 0.00 (NA) — Standard deviation does not apply when n = 1. | 7.14 (11.202)
  Endocrine, EOT up to week 82: number analyzed (Participants) | 41 | 76
  Endocrine, EOT up to week 82 | 9.49 (15.627) | 15.20 (18.755)
  G.I., Baseline: number analyzed (Participants) | 65 | 111
  G.I., Baseline | 23.69 (20.183) | 26.19 (21.328)
  G.I., week 4: number analyzed (Participants) | 53 | 99
  G.I., week 4 | 23.02 (20.488) | 23.39 (18.958)
  G.I., week 8: number analyzed (Participants) | 34 | 89
  G.I., week 8 | 22.34 (18.398) | 27.53 (21.341)
  G.I., week 20: number analyzed (Participants) | 8 | 56
  G.I., week 20 | 25.63 (14.056) | 22.31 (18.837)
  G.I., week 32: number analyzed (Participants) | 4 | 38
  G.I., week 32 | 25.00 (11.386) | 26.84 (19.879)
  G.I., week 44: number analyzed (Participants) | 1 | 14
  G.I., week 44 | 0.00 (NA) — Standard deviation does not apply when n = 1. | 20.95 (16.714)
  G.I., EOT up to week 82: number analyzed (Participants) | 41 | 76
  G.I., EOT up to week 82 | 25.85 (19.899) | 30.48 (24.484)
  Treatment, baseline: number analyzed (Participants) | 33 | 69
  Treatment, baseline | 9.26 (11.675) | 18.44 (19.374)
  Treatment, week 4: number analyzed (Participants) | 42 | 84
  Treatment, week 4 | 17.72 (15.337) | 22.22 (20.077)
  Treatment, week 8: number analyzed (Participants) | 23 | 77
  Treatment, week 8 | 16.18 (19.528) | 20.27 (17.283)
  Treatment, week 20: number analyzed (Participants) | 6 | 47
  Treatment, week 20 | 28.70 (21.493) | 19.74 (19.755)
  Treatment, week 32: number analyzed (Participants) | 2 | 27
  Treatment, week 32 | 27.78 (7.857) | 24.49 (23.684)
  Treatment, week 44: number analyzed (Participants) | 1 | 11
  Treatment, week 44 | 16.67 (NA) — Standard deviation does not apply when n = 1. | 18.18 (18.936)
  Treatment, EOT up to week 82: number analyzed (Participants) | 35 | 58
  Treatment, EOT up to week 82 | 22.06 (21.705) | 24.81 (21.735)
  Social function, Baseline: number analyzed (Participants) | 66 | 110
  Social function, Baseline | 39.56 (23.721) | 47.42 (25.726)
  Social function, week 4: number analyzed (Participants) | 54 | 100
  Social function, week 4 | 36.52 (26.294) | 45.28 (27.483)
  Social function, week 8: number analyzed (Participants) | 31 | 87
  Social function, week 8 | 38.35 (23.629) | 46.49 (26.265)
  Social function, week 20: number analyzed (Participants) | 8 | 56
  Social function, week 20 | 40.28 (14.472) | 42.66 (25.648)
  Social function, week 32: number analyzed (Participants) | 4 | 38
  Social function, week 32 | 38.89 (14.344) | 48.54 (23.735)
  Social function, week 44: number analyzed (Participants) | 1 | 14
  Social function, week 44 | 33.33 (NA) — Standard deviation does not apply when n = 1. | 40.08 (26.165)
  Social function, EOT up to week 82: number analyzed (Participants) | 43 | 75
  Social function, EOT up to week 82 | 38.89 (25.051) | 54.22 (28.428)
  Disease-related worries, Baseline: number analyzed (Participants) | 66 | 110
  Disease-related worries, Baseline | 43.10 (25.599) | 53.94 (27.664)
  Disease-related worries, week 4: number analyzed (Participants) | 54 | 100
  Disease-related worries, week 4 | 39.20 (28.562) | 46.33 (28.165)
  Disease-related worries, week 8: number analyzed (Participants) | 30 | 87
  Disease-related worries, week 8 | 40.56 (28.183) | 47.32 (28.541)
  Disease-related worries, week 20: number analyzed (Participants) | 8 | 56
  Disease-related worries, week 20 | 37.50 (8.267) | 46.83 (32.096)
  Disease-related worries, week 32: number analyzed (Participants) | 4 | 38
  Disease-related worries, week 32 | 38.89 (11.111) | 53.51 (27.137)
  Disease-related worries, week 44: number analyzed (Participants) | 1 | 14
  Disease-related worries, week 44 | 33.33 (NA) — Standard deviation does not apply when n=1. | 44.05 (32.647)
  Disease-related worries, EOT up to week 82: number analyzed (Participants) | 43 | 75
  Disease-related worries, EOT up to week 82 | 42.89 (28.876) | 55.04 (31.667)
  Muscle/bone pain, Baseline: number analyzed (Participants) | 65 | 109
  Muscle/bone pain, Baseline | 26.67 (33.347) | 29.66 (31.210)
  Muscle/bone pain, week 4: number analyzed (Participants) | 54 | 100
  Muscle/bone pain, week 4 | 24.07 (29.966) | 33.00 (31.956)
  Muscle/bone pain, week 8: number analyzed (Participants) | 31 | 88
  Muscle/bone pain, week 8 | 31.18 (34.357) | 33.33 (33.524)
  Muscle/bone pain, week 20: number analyzed (Participants) | 8 | 56
  Muscle/bone pain, week 20 | 41.67 (15.430) | 34.52 (33.614)
  Muscle/bone pain, week 32: number analyzed (Participants) | 4 | 38
  Muscle/bone pain, week 32 | 50.00 (19.245) | 40.35 (34.795)
  Muscle/bone pain, week 44: number analyzed (Participants) | 1 | 14
  Muscle/bone pain, week 44 | 33.33 (NA) — Standard deviation does not apply when n=1. | 26.19 (26.726)
  Muscle/bone pain, EOT up to week 82: number analyzed (Participants) | 42 | 75
  Muscle/bone pain, EOT up to week 82 | 34.13 (28.973) | 40.89 (33.141)
  Sexual function, Baseline: number analyzed (Participants) | 47 | 78
  Sexual function, Baseline | 35.46 (32.899) | 39.32 (40.468)
  Sexual function, week 4: number analyzed (Participants) | 38 | 75
  Sexual function, week 4 | 21.05 (26.191) | 40.89 (40.483)
  Sexual function, week 8: number analyzed (Participants) | 22 | 63
  Sexual function, week 8 | 28.79 (33.007) | 43.92 (40.083)
  Sexual function, week 20: number analyzed (Participants) | 3 | 35
  Sexual function, week 20 | 33.33 (33.333) | 38.10 (39.724)
  Sexual function, week 32: number analyzed (Participants) | 3 | 24
  Sexual function, week 32 | 11.11 (19.245) | 29.17 (35.864)
  Sexual function, week 44: number analyzed (Participants) | 0 | 7
  Sexual function, week 44 |  | 47.62 (46.576)
  Sexual function, EOT up to week 82: number analyzed (Participants) | 31 | 47
  Sexual function, EOT up to week 82 | 25.81 (28.166) | 48.94 (43.323)
  Communication function, Baseline: number analyzed (Participants) | 66 | 108
  Communication function, Baseline | 7.58 (16.325) | 9.88 (22.904)
  Communication function, week 4: number analyzed (Participants) | 53 | 98
  Communication function, week 4 | 8.18 (17.179) | 6.46 (15.626)
  Communication function, week 8: number analyzed (Participants) | 30 | 86
  Communication function, week 8 | 12.22 (18.535) | 9.69 (19.714)
  Communication function, week 20: number analyzed (Participants) | 7 | 55
  Communication function, week 20 | 14.29 (17.817) | 10.30 (19.108)
  Communication function, week 32: number analyzed (Participants) | 4 | 38
  Communication function, week 32 | 8.33 (16.667) | 7.89 (19.658)
  Communication function, week 44: number analyzed (Participants) | 1 | 14
  Communication function, week 44 | 0.00 (NA) — Standard deviation does not apply when n=1. | 4.76 (12.105)
  Communication function, EOT up to week 82: number analyzed (Participants) | 42 | 74
  Communication function, EOT up to week 82 | 12.70 (22.028) | 12.61 (23.214)
  Body image, Baseline: number analyzed (Participants) | 65 | 107
  Body image, Baseline | 15.90 (28.932) | 22.43 (34.195)
  Body image, week 4: number analyzed (Participants) | 53 | 98
  Body image, week 4 | 15.09 (27.399) | 22.79 (31.239)
  Body image, week 8: number analyzed (Participants) | 31 | 83
  Body image, week 8 | 21.51 (27.953) | 26.10 (31.256)
  Body image, week 20: number analyzed (Participants) | 8 | 55
  Body image, week 20 | 16.67 (17.817) | 30.30 (34.708)
  Body image, week 32: number analyzed (Participants) | 4 | 37
  Body image, week 32 | 0.00 (0.000) | 28.83 (33.483)
  Body image, week 44: number analyzed (Participants) | 1 | 14
  Body image, week 44 | 0.00 (NA) — Standard deviation does not apply when n=1. | 30.95 (27.625)
  Body image, EOT up to week 82: number analyzed (Participants) | 42 | 73
  Body image, EOT up to week 82 | 23.02 (32.500) | 34.70 (37.449)

6. Secondary Outcome: Number and Percentage of Participants With Ratings of 'no Problem, 'Some Problem' and 'Extreme Problem' in the EuroQol Five Dimensions Questionnaire (EQ-5D) (Core)
Description: The EQ-5D is divided into two distinct sections. The first section includes one item addressing each of five dimensions (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression). Patients rate each of these items from "no problem," "some problem," or "extreme problem." A composite health index is then defined by combining the levels for each dimension. The second section of the questionnaire measures self-rated (global) health status utilizing a vertically oriented visual analogue scale where 100 represents the "best possible health state" and 0 represents the "worst possible health state." Respondents are asked to rate their current health by placing a mark along this continuum. The scores from each section are then transformed into a single health utility score. Overall scores range from 0 to 1 with lower scores representing a higher level of dysfunction.
Time Frame: Baseline, weeks 4, 8, 20, 32, 44, and end of treatment (EOT) up to week 82
Population: The full analysis set, which consisted of all participants who received at least one dose of everolimus, was analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- pNET (Core); Non-pNET (Core): Participants received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 126 | 120
Participants
  Baseline, Mobility, No problem | 84 | 76
  Baseline, Mobility, Some problem | 31 | 35
  Baseline, Mobility, Extreme problem | 2 | 1
  Baseline, Self-care, No problem | 100 | 102
  Baseline, Self-care, Some problem | 15 | 10
  Baseline, Self-care, Extreme problem: number analyzed (Participants) | 126 | 0
  Baseline, Self-care, Extreme problem | 2 |
  Baseline, Usual activities, No problem | 71 | 60
  Baseline, Usual activities, Some problem | 43 | 46
  Baseline, Usual actvities, Extreme problem | 4 | 6
  Baseline, Pain/Discomfort, No problem | 59 | 40
  Baseline, Pain/discomfort, Some problem | 52 | 66
  Baseline, Pain/discomfort, Extreme problem | 6 | 7
  Baseline, Anxiety/depression, No problem | 65 | 53
  Baseline, Anxiety/depression, Some problem | 47 | 54
  Baseline, Anxiety/depression, Extreme problem | 5 | 6
  Week 4, Mobility, No problem | 72 | 66
  Week 4, Mobility, Some problem | 27 | 37
  Week 4, Mobility, Extreme problem | 2 | 1
  Week 4, Self-care, No problem | 89 | 86
  Week 4, Self-care, Some problem | 10 | 16
  Week 4, Self-care, Extreme problem | 3 | 2
  Week 4, Usual activities, No problem | 66 | 55
  Week 4, Usual activities, Some problem | 31 | 42
  Week 4, Usual activities, Extreme problem | 4 | 7
  Week 4, Pain/discomfort, No problem | 39 | 30
  Week 4, Pain/discomfort, Some problem | 58 | 64
  Week 4, Pain/discomfort, Extreme problem | 3 | 8
  Week 4, Anxiety/depression, No problem | 54 | 57
  Week 4, Anxiety depression, Some problem | 46 | 43
  Week 4, Anxiety/depression, Extreme problem | 1 | 3
  Week 8, Mobility, No problem | 48 | 45
  Week 8, Mobility, Some problem | 24 | 37
  Week 8, Mobility, Extreme problem | 2 | 3
  Week 8, Self-care, No problem | 61 | 70
  Week 8, Self-care, Some problem | 7 | 15
  Week 8, Self-care, Extreme problem | 6 | 1
  Week 8, Usual activities, No problem | 46 | 40
  Week 8, Usual activities, Some problem | 23 | 41
  Week 8, Usual activties, Extreme problem | 4 | 5
  Week 8, Pain/discomfort, No problem | 34 | 25
  Week 8, Pain/discomfort, Some problem | 32 | 52
  Week 8, Pain/discomfort, Extreme problem | 7 | 10
  Week 8, Anxiety/depression, No problem | 43 | 38
  Week 8, Anxiety/depression, Some problem | 30 | 41
  Week 8, Anxiety/depression, Extreme problem | 1 | 8
  Week 20, Mobility, No problem | 26 | 37
  Week 20, Mobility, Some problem | 3 | 17
  Week 20, Mobility, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 20, Mobility, Extreme problem |  | 1
  Week 20, Self-care, No problem | 25 | 49
  Week 20, Self-care, Some problem | 4 | 6
  Week 20, Self-care, Extreme problem: number analyzed (Participants) | 0 | 0
  Week 20, Usual activities, No problem | 18 | 30
  Week 20 Usual activities, Some problem | 10 | 22
  Week 20, Usual activities, Extreme problem | 1 | 2
  Week 20, Pain/discomfort, No problem | 12 | 19
  Week 20, Pain/discomfort, Some problem | 16 | 34
  Week 20, Pain/discomfort, Extreme problem | 1 | 2
  Week 20, Anxiety/depression, No problem | 16 | 27
  Week 20, Anxiety/depression, Some problem | 12 | 23
  Week 20, Anxiety/depression, Extreme problem | 1 | 5
  Week 32, Mobility, No problem | 3 | 25
  Week 32, Mobility, Some problem | 2 | 12
  Week 32, Mobility, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 32, Mobility, Extreme problem |  | 2
  Week 32, Self-care, No problem | 5 | 32
  Week 32, Self-care, Some problem: number analyzed (Participants) | 0 | 120
  Week 32, Self-care, Some problem |  | 3
  Week 32, Self-care, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 32, Self-care, Extreme problem |  | 2
  Week 32, Usual activities, No problem | 4 | 22
  Week 32, Usual activities, Some problem | 1 | 14
  Week 32, Usual activities, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 32, Usual activities, Extreme problem |  | 3
  Week 32, Pain/discomfort, No problem | 1 | 10
  Week 32, Pain/discomfort, Some problem | 4 | 27
  Week 32, Pain/discomfort, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 32, Pain/discomfort, Extreme problem |  | 2
  Week 32, Anxiety/depression, No problem | 4 | 20
  Week 32, Anxiety/depression, Some problem | 1 | 14
  Week 32, Anxiety/depression, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 32, Anxiety/depression, Extreme problem |  | 5
  Week 44, Mobility, No problem | 2 | 9
  Week 44, Mobility, Some problem | 1 | 4
  Week 44, Mobility, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 44, Mobility, Extreme problem |  | 1
  Week 44, Self-care, No problem | 3 | 12
  Week 44, Self-care, Some problem: number analyzed (Participants) | 0 | 120
  Week 44, Self-care, Some problem |  | 2
  Week 44, Self-care, Extreme problem: number analyzed (Participants) | 0 | 0
  Week 44, Usual activities, No problem: number analyzed (Participants) | 0 | 120
  Week 44, Usual activities, No problem |  | 6
  Week 44, usual activities, Some problem | 3 | 7
  Week 44, usual activities, Extreme problem: number analyzed (Participants) | 0 | 0
  Week 44, Pain/discomfort, No problem: number analyzed (Participants) | 0 | 120
  Week 44, Pain/discomfort, No problem |  | 6
  Week 44, Pain/discomfort, Some problem | 3 | 8
  Week 44, Pain/discomfort, Extreme problem: number analyzed (Participants) | 0 | 0
  Week 44, Anxiry/depression, No problem | 1 | 7
  Week 44, Anxiety/depression, Some problem | 2 | 6
  Week 44, Anxiety/depression, Extreme problem: number analyzed (Participants) | 0 | 120
  Week 44, Anxiety/depression, Extreme problem |  | 1
  EOT up to Week 82, Mobility, No problem | 59 | 42
  EOT up to Week 82, Mobility, Some problem | 23 | 31
  EOT up to Week 82, Mobility, Extreme problem | 4 | 4
  EOT up to Week 82, Self-care, No problem | 69 | 56
  EOT up to Week 82, Self-care, Some problem | 12 | 19
  EOT up to Week 82, Self-care, Extreme problem | 2 | 1
  EOT up toWeek 82, Usual activities, No problem | 54 | 29
  EOT up to Week 82, Usual activities, Some problem | 24 | 36
  EOT up to Week 82, Usual activities, Extreme prob. | 5 | 11
  EOT up to Week 82, Pain/discomfort, No problem | 43 | 18
  EOT up to Week 82, Pain/discomfort, Some problem | 36 | 48
  EOT up to Week 82, Pain/discomfort, Extreme prob. | 5 | 11
  EOT up to Week 82, Anxiety/depression, No problem | 48 | 31
  EOT up to Week 82, Anxiety/depression, Some prob. | 33 | 40
  EOT up toWeek 82, Anxiety/depression, Extreme prob | 3 | 6

7. Secondary Outcome: Mean EQ-5D Visual Analogue Scale (VAS) Score (Core)
Description: as for outcome 6
Time Frame: Baseline, weeks 4, 8, 20, 32, 44, and end of treatment (EOT) up to week 82
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 126 | 120
units on a scale
  Baseline: number analyzed (Participants) | 118 | 111
  Baseline | 68.8 (19.90) | 63.9 (19.09)
  Week 4: number analyzed (Participants) | 100 | 104
  Week 4 | 69.3 (18.06) | 63.8 (18.78)
  Week 8: number analyzed (Participants) | 73 | 88
  Week 8 | 64.6 (21.77) | 61.2 (18.65)
  Week 20: number analyzed (Participants) | 28 | 54
  Week 20 | 67.4 (19.58) | 64.6 (15.51)
  Week 32: number analyzed (Participants) | 5 | 37
  Week 32 | 42.6 (24.67) | 62.0 (17.65)
  Week 44: number analyzed (Participants) | 3 | 13
  Week 44 | 66.7 (15.28) | 68.6 (18.71)
  EOT up to Week 82: number analyzed (Participants) | 86 | 76
  EOT up to Week 82 | 66.5 (20.64) | 55.3 (23.02)

8. Secondary Outcome: Investigator-assessed Best Overall Response (Core)
Description: Best overall response was determined from the sequence of investigator overall lesions responses according to Response Evaluation Criteria in Solid Tumors (RECIST). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Progression, a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from the start of treatment, every 12 weeks for the first year and then every 6 months up to 19 months
Population: The full analysis set, which consisted of all participants who received at least one dose, was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | pNET (Core) | Non-pNET (Core)
Number analyzed (Participants) | 126 | 120
Participants
  Partial response (PR) | 2 | 1
  Stable disease (SD) | 74 | 84
  Progressive disease (PD) | 9 | 8
  Unknown | 41 | 27
  Objective response rate (complete response or PR) | 2 | 1

9. Secondary Outcome: Investigator-assessed Progression Free Survival (PFS) (E1)
Description: PFS was defined as the time from the date of the start of therapy in the extension study to the date of the first radiologically documented disease progression or death due to any cause. If a participant had not progressed or died at the analysis cut-off date or when he/she received any further anti-neoplastic therapy, PFS was censored at the time of the last adequate tumor evaluation before the cut-off date or the anti-neoplastic therapy start date.
Time Frame: from first date of treatment in the extension up to 4 years
Population: The full analysis set, which consisted of all participants who received at least one dose of everolimus during the extension, was analyzed
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Lung NET (E1); GI NET (E1): Participants received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
Arm/Group | Lung NET (E1) | GI NET (E1)
Number analyzed (Participants) | 4 | 11
Days | 159 [10 to 1074] | 655 [9 to NA] — The upper limit of the 95% confidence interval was not estimable since there were too few number of participants at this time point.

10. Secondary Outcome: Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) Score at the End of Treatment From Baseline (Baseline = First Day of Treatment in the Extension) (E1)
Description: The EORTC QLQ-C30 contains 30 questions assessed by the participant. There are 9 multiple-item scales: 5 scales that assess aspects of functioning (physical, role, cognitive, emotional, and social); 3 symptom scales (Fatigue, Pain, and Nausea and Vomiting); and a global health status and QOL scale. There are 5 single-item measures assessing additional symptoms (i.e., dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and a single item concerning perceived financial impact of the disease. All but two questions have 4-point scales ranging from "Not at all" to "Very much." The two questions concerning global health status and QOL have 7 point scales with ratings ranging from "Very poor" to "Excellent." For each of the 14 domains, changes are calculated as value at later time point minus value at baseline, and final scores are transformed such that they range from 0-100, where higher scores indicate better outcomes. A positive change from baseline indicates improvement.
Time Frame: baseline, every 12 weeks and up to 4 years
Population: Only participants from the full analysis set, who had both baseline and end of treatment measurements, were included in the analysis. The full analysis set, which consisted of all participants who received at least one dose of everolimus during the extension, was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GI NET: Participants received Everolimus 10 mg orally once daily until documented tumor progression, unacceptable toxicity or any other reason.
Arm/Group | Lung NET (E1) | GI NET
Number analyzed (Participants) | 1 | 6
score on a scale
  Global health status/QoL | 0.00 (NA) — Standard deviation does not apply when n=1. | -0.00 (11.785)
  Functional scale: Physical functioning | 6.67 (NA) — Standard deviation does not apply when n=1. | 0.00 (7.303)
  Functional scale: Role functioning | -16.67 (NA) — Standard deviation does not apply when n=1. | 5.56 (22.771)
  Functional scale: Emotional functioning | -25.00 (NA) — Standard deviation does not apply when n=1. | -1.85 (17.003)
  Functional scale: Cognitive functioning | -66.67 (NA) — Standard deviation does not apply when n=1. | -16.67 (21.082)
  Functional scale: Social functioning | 0.00 (NA) — Standard deviation does not apply when n=1. | -8.33 (9.129)
  Symptom scale: Fatigue | 0.00 (NA) — Standard deviation does not apply when n=1. | -3.70 (22.951)
  Symptom scale: Nausea and vomiting | 0.00 (NA) — Standard deviation does not apply when n=1. | 0.00 (18.257)
  Symptom scale: Pain | 0.00 (NA) — Standard deviation does not apply when n=1. | 16.67 (27.889)
  Symptom scale: Dyspnea | 0.00 (NA) — Standard deviation does not apply when n=1. | -5.56 (13.608)
  Symptom scale: Insomnia | 33.33 (NA) — Standard deviation does not apply when n=1. | 11.11 (17.213)
  Symptom scale: Appetite loss | 0.00 (NA) — Standard deviation does not apply when n=1. | 0.00 (21.082)
  Symptom scale: Constipation | 0.00 (NA) — Standard deviation does not apply when n=1. | 5.56 (25.092)
  Symptom scale: Diarrhea | 0.00 (NA) — Standard deviation does not apply when n=1. | -16.67 (45.947)
  Symptom scale: Financial difficulties | -33.33 (NA) — Standard deviation does not apply when n=1. | 16.67 (18.257)

11. Secondary Outcome: Change in EORTC QLQ-G.I. NET21 Score at the End of Treatment From Baseline (Baseline = First Day of Treatment in the Extension) (E1)
Description: The EORTC QLQ-G.I. NET21 contains 21 questions and has three defined multi-item symptom scales (endocrine - 3 questions, gastrointestinal - 5 questions, and treatment related side effects - 3 questions), two single item symptoms (bone/muscle pain and concern about weight loss), two psychosocial scales (social function - 3 questions, disease-related worries - 3 questions) and two other single items (sexuality and communication). For each of the 9 domains, final scores are transformed such that they range from 0-100, where higher scores indicate worsening outcomes. A positive change from baseline indicates worsening.
Time Frame: baseline, every 12 weeks and up to 4 years
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung NET (E1) | GI NET
Number analyzed (Participants) | 4 | 11
units on a scale
  Social function: number analyzed (Participants) | 1 | 6
  Social function | 11.11 (NA) — Standard deviation does not apply when n=1. | 7.41 (22.951)
  Disease-related worries: number analyzed (Participants) | 1 | 6
  Disease-related worries | 44.44 (NA) — Standard deviation does not apply when n=1. | -0.93 (7.384)
  Sexual function: number analyzed (Participants) | 0 | 1
  Sexual function |  | 50.00 (43.033)
  Communicative functioning: number analyzed (Participants) | 1 | 6
  Communicative functioning | 0.00 (NA) — Standard deviation does not apply when n=1. | 11.11 (17.213)
  Endocrine scale: number analyzed (Participants) | 1 | 6
  Endocrine scale | 11.11 (NA) — Standard deviation does not apply when n=1. | 5.56 (18.257)
  G.I. scale: number analyzed (Participants) | 1 | 6
  G.I. scale | 0.00 (NA) — Standard deviation does not apply when n=1. | 14.44 (23.633)
  Treatment scale: number analyzed (Participants) | 1 | 5
  Treatment scale | -16.67 (NA) — Standard deviation does not apply when n=1. | 5.56 (12.423)
  Muscle/bone pain symptom: number analyzed (Participants) | 0 | 6
  Muscle/bone pain symptom |  | 33.33 (29.814)
  Body image: number analyzed (Participants) | 1 | 6
  Body image | 0.00 (NA) — Standard deviation does not apply when n=1. | 0.00 (21.082)

12. Secondary Outcome: Change in EuroQol Five Dimensions Questionnaire (EQ-5D) Score at the End of Treatment From Baseline (Baseline = First Day of Treatment in the Extension) (E1)
Description: The EQ-5D contains 2 sections:1st section has 1 item addressing each of 5 dimensions (mobility, self-care, usual activity, pain/discomfort, anxiety/depression). Each dimension has 3 levels: no problems, some problems, extreme problems, 1-3, respectively. A health state is defined by combining 1 level from each dimension. 243 health states are possible. Each state is referred to in a 5 digit code. E.g., state 11111 indicates no problems on any dimension, while state 11223 indicates no problems with mobility and self-care, some problems with performing usual activities, moderate pain or discomfort and extreme anxiety or depression. The 2nd section measures self-rated health status using a visual analogue scale (VAS) where 100 represents best possible health and 0 represents worst possible health. Patients are asked to rate their current health by placing a mark on the VAS. Scores from each section are then transformed into an overall score of 0 or 1, with 0= higher level of dysfunction.
Time Frame: baseline, every 12 weeks and up to 4 years
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung NET (E1) | GI NET
Number analyzed (Participants) | 1 | 6
units on a scale
  Composite health index | 7.26 (NA) — Standard deviation does not apply when n=1. | -8.58 (13.302)
  Self-rated health status | -10.00 (NA) — Standard deviation does not apply when n=1. | -4.17 (21.479)

13. Secondary Outcome: Investigator-assessed Best Overall Response During the Extension Phase (E1)
Description: as for outcome 8
Time Frame: from the start of treatment, every 12 weeks for the first year and then every 6 months up to 4 years
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Lung NET (E1) | GI NET
Number analyzed (Participants) | 4 | 11
Participants
  Complete response | 0 | 0
  Partial response | 0 | 1
  Stable disease | 2 | 7
  Progressive disease | 2 | 3
  Unknown | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 19 month for the core and up to 4 years for the extension
Groups:
- pNET (Core): pNET (Core)
- Non-pNET (Core): Non-pNET (Core)
- Lung NET (E1): Lung NET (E1)
- GI NET (E1): GI NET (E1)
Arm/Group | pNET (Core) | Non-pNET (Core) | Lung NET (E1) | GI NET (E1)
Serious Adverse Events (participants affected / at risk) | 25/123 | 59/117 | 1/4 | 4/11
Other Adverse Events (participants affected / at risk) | 73/123 | 89/117 | 4/4 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | pNET (Core) (N=123) | Non-pNET (Core) (N=117) | Lung NET (E1) (N=4) | GI NET (E1) (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Retinal vascular thrombosis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Device occlusion (General disorders) | 1 | 0 | 0 | 0
Euthanasia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 5 | 0 | 0
General physical health deterioration (General disorders) | 2 | 7 | 0 | 1
Impaired healing (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 2 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 6 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Antineutrophil cytoplasmic antibody increased (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 1
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 2 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | pNET (Core) (N=123) | Non-pNET (Core) (N=117) | Lung NET (E1) (N=4) | GI NET (E1) (N=11)
Anaemia (Blood and lymphatic system disorders) | 7 | 10 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 5 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 10 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 10 | 34 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 10 | 10 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 11 | 13 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 5 | 1 | 0
Asthenia (General disorders) | 12 | 6 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 13 | 0 | 3
Generalised oedema (General disorders) | 1 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 12 | 5 | 0 | 0
Oedema (General disorders) | 1 | 3 | 1 | 0
Oedema peripheral (General disorders) | 5 | 15 | 0 | 4
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 8 | 5 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 2
Erysipelas (Infections and infestations) | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 2
Laryngitis (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 2 | 5
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 3 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 4 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 5 | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 3 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 9 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 5 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 6 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 9 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 3 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 0 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 5 | 6 | 0 | 5
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.